CLINICAL TRIAL: NCT07210944
Title: Research Protocol for a Randomized Controlled Trial on Brain Network Study of Upper Limb Motor Dysfunction in Stroke Patients Treated With Scalp Acupuncture Combined With rTMS
Brief Title: Scalp Acupuncture Combined With rTMS for Upper Limb Motor Dysfunction in Stroke: A Brain Network Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Debiao Kong (Other)
Responsible Party: Sponsor-Investigator, Debiao Kong, resident physician, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZSLL-KY-2025-046
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Upper Extremity; Acupuncture Therapy; Stroke; Transcranial Magnetic Stimulation Repetitive; Motor Disorders
Keywords: Conventional rehabilitation therapy; Scalp Acupuncture; Upper Limb; Repetitive Transcranial Magnetic Stimulation; Motor Disorders
MeSH Terms: conditions — Stroke; Motor Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Repeat transcranial magnetic stimulation and conventional treatment
  Interventions: Device: Repetitive transcranial magnetic stimulation; Combination Product: Conventional rehabilitation treatment
- experimental group (Experimental): Repeat transcranial magnetic stimulation and scalp acupuncture and conventional treatment
  Interventions: Device: Repetitive transcranial magnetic stimulation; Procedure: Scalp acupuncture; Combination Product: Conventional rehabilitation treatment

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Transcranial magnetic stimulation applied a figure-8 coil to the premotor area at 80%-100% of the healthy-side MEP threshold. Treatment lasted 20 min in two phases: weeks 1-2 on the ipsilateral M1 (1Hz, 10s on/5s off), and weeks 3-4 on the contralateral M1 (10Hz, 3s on/12s off). Treat once a day, 5 days a week, for a total of 4 weeks.
Procedure: Scalp acupuncture — Scalp acupuncture selected bilateral upper-limb cortical MEP points (2 points total). The healthy-side hot spot was identified first; if the affected side had no MEP, its mirror point was used. Needles were inserted from point A (affected) to B (healthy) and beyond along the AB line. After insertion, needles were rotated for 2-3 min, manipulated every 10 min, and retained for 30 min. Treat once a day, 5 days a week, for a total of 4 weeks.
  Arms: experimental group
Combination Product: Conventional rehabilitation treatment — Conventional drug therapy included secondary stroke prevention, neurotrophy, and improved cerebral circulation. Routine rehabilitation involved exercise, occupational, and physical therapies, with a total daily treatment time of 90 minutes.

SUMMARY:
This study aims to compare the improvement effects of the rTMS (repetitive transcranial magnetic stimulation) combined with conventional rehabilitation therapy group with the rTMS combined with scalp acupuncture and conventional rehabilitation therapy group. Through statistical analysis of the results obtained from functional near-infrared spectroscopy technology during task states, the investigators elucidate the neuroregulatory mechanism of scalp acupuncture combined with rTMS in improving upper limb motor function in stroke patients under MEP localization, and provide evidence for a more optimal rehabilitation program for post-stroke upper limb motor dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for stroke (symptoms and signs, imaging indicators, etc.), and are independently diagnosed by two deputy chief physicians
* Age 18-70 years old, first episode, duration 1-6 months
* The diagnostic criteria for upper limb dysfunction align with the Brunnstrom staging system: patients in Brunnstrom stages II to IV. Stage II: patients exhibit associative responses and can perform coordinated movements, with minimal voluntary movements; Stage III: patients show voluntary coordinated movements, such as grasping with the hand but not extending; Stage IV: patients can perform isolated movements, such as pinching with the hand and limited extension
* No severe visual or hearing impairment, able to cooperate with relevant assessments and tests
* The score of the Mini-Mental State Examination is ≥20 points
* Vital signs are stable, with no signs of progressive neurological symptoms
* The patient or legal guardian agrees and signs the informed consent form

Exclusion Criteria:

* Severe visual impairment, hemispatial neglect, body image disorder
* Individuals who cannot undergo rTMS treatment due to reasons such as metal implants, cardiac pacemakers, or skull defects
* Previous history of brain tumor, brain trauma, epilepsy, and risk of epileptic seizures
* Any other factors that affect assessment and treatment
* Dysfunction of limb movement caused by other reasons (such as trauma, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Maximum amplitude of motor evoked potential | One day before treatment, four weeks after treatment
  It refers to the potential difference between the peak and trough of the motor evoked potential, reflecting the excitability of the cerebral cortex and neural pathways. It is detected using an RD-CCY type TMS stimulator in conjunction with a Viking Quest 4-channel surface electromyography recorder from the American company Neuropad.
Fugl-Meyer Assessment-Upper Extremities | One day before treatment, four weeks after treatment
  It is a widely used standardized assessment tool in the rehabilitation of upper limb motor dysfunction after stroke. The FMA divides upper limb motor function into multiple dimensions, including reflex activity, coordinated movement, isolated movement, wrist and hand function, through systematic scoring items. A total of 33 items are included. Each item is scored on a 3-point scale (0-2 points), with a total score of 66 (upper limb part). Higher scores indicate better recovery of upper limb motor function.

SECONDARY OUTCOMES:
Action Research Arm Test | One day before treatment, four weeks after treatment
  It includes 4 parts: grasping, holding, pinching, and gross motor function, with a total of 19 items. Each item is scored on a 4-point scale (0-3 points), with a total of 57 points. The higher the score, the better the recovery of upper limb motor function.
Modified Barthel Index | One day before treatment, four weeks after treatment
  It is used to assess patients' ability to perform activities of daily living. It includes 10 items: eating, dressing, using the toilet, defecating, urinating, grooming, bathing, climbing stairs, transferring, and walking. The total score ranges from 0 to 100, with higher scores indicating better ability to perform activities of daily living. A score of >60 indicates that the patient can live independently.
Functional near-infrared spectroscopy | One day before treatment, two weeks after treatment, four weeks after treatment
  Data were collected using a 35-channel fNIRS imaging device, NirSmart (HuiChuang, China), during resting state and scalp acupuncture stimulation. The device includes 17 light source probes and 14 detection probes, forming 35 effective channels in the experimental design, covering the forehead, bilateral frontal lobes, and motor areas. Continuous wave, near-infrared wavelength (760-850nm) signals were used with a sampling frequency of 11Hz, allowing real-time and effective monitoring of changes in the concentration of oxyhemoglobin and deoxyhemoglobin in the healthy side of the subject's brain. Based on coordinate information, the 35 channels were divided into five regions of interest in the left and right cerebral cortexes of the subject, namely the bilateral motor area, bilateral temporal lobe and forehead.

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No